CLINICAL TRIAL: NCT03823326
Title: Paediatric Oximetry Algorithms - Normative Data Collection
Status: Completed | Type: Observational
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SCH-2155
Record Dates: First submitted 2019-01-25; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Sleep Apnea Syndromes in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To undertake normative data collection of existing clinical algorithms using existing oximetry technology.

DETAILED DESCRIPTION:
Paediatric patients who are undergoing routine diagnostic pulse oximetry, will be approached to also wear an additional oximeter at the same time so that comparisons between two oximeters and their clinical algorithms can be compared.

ELIGIBILITY:
Inclusion Criteria:

* All children who have been referred for a clinical overnight pulse oximetry test

Exclusion Criteria:

* Families who do not understand written English if an interpreter is not present for clinical reasons
* Times when the kit is already being used for another recruit
* If children do not attend with the legal guardian and so informed consent cannot be signed
* Patient is deemed too unwell by clinical team to be approached about the research

Ages: 1 Month to 16 Years | Sex: All
Age Groups: Child
Study Population: All children aged 1 month - 16 years who are undergoing an overnight pulse oximetry investigation.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Oximetry Raw data | Overnight (8-10 hours) of pulse oximetry data is collected from participants and then they have completed the study. It is a single time frame of data collection.
  2 second data dumps of SpO2 signals from an overnight trace
Pulse Rate Raw data | Overnight (8-10 hours) of pulse oximetry data is collected from participants and then they have completed the study. It is a single time frame of data collection
  2 second data dumps of SpO2 signals from an overnight trace

OTHER OUTCOMES:
Age | Taken at time of consent
  Age of child at time of oximetry
Gender | Taken at time of consent
  Gender of child

CONTACTS AND LOCATIONS:
Overall Officials: Heather E Elphick, MbChBMDMRCPH, Principal Investigator — Sheffield Children's Hospital
Locations (1):
- Clinical Research Facility, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No